CLINICAL TRIAL: NCT02944825
Title: A Randomized, Prospective, Single-Blinded Control Trial to Assess the Need for Antibiotic Prophylaxis With Routine Ureteral Stent Removal After Kidney Stone Procedure
Brief Title: Antibiotic Prophylaxis With Routine Ureteral Stent Removal
Acronym: STENTABX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Genesis HealthCare (Other)
Responsible Party: Principal Investigator, Roger L Sur, M.D., Director of Endourology, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 160160
Record Dates: First submitted 2016-10-24; First posted 2016-10-26 (Estimated); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Urolithiasis; UTI
Keywords: Urolithiasis; UTI
MeSH Terms: conditions — Urolithiasis | interventions — Ciprofloxacin; Trimethoprim, Sulfamethoxazole Drug Combination

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Antibiotic (Active Comparator): Patients randomized to the intervention arm will be provided a single oral dose of prophylactic oral antibiotic at the time of cystoscopic stent removal
  Interventions: Drug: Ciprofloxacin; Drug: trimethoprim/sulfamethoxazole
- No Antibiotic (Active Comparator): Patients randomized to the non-intervention arm will not undergo prophylaxis at the time of cystoscopic stent removal
  Interventions: Drug: No Intervention

INTERVENTIONS:
Drug: Ciprofloxacin — first line prophylactic oral antibiotic
  Arms: Antibiotic
Drug: trimethoprim/sulfamethoxazole — second line prophylactic oral antibiotic
  Other Names: Bactrim; Septra
  Arms: Antibiotic
Drug: No Intervention — No intervention
  Arms: No Antibiotic

SUMMARY:
This study will be a single-institutional randomized, single-blinded prospectively controlled clinical trial of a single dose of Ciprofloxicin 500mg antibiotic tablet as prophylaxis at the time of office flexible cystoscopy with ureteral stent removal. The control group will be no prophylaxis oral antibiotics.

DETAILED DESCRIPTION:
This study will be a single-institutional randomized, single-blinded prospectively controlled clinical trial of a single dose of Ciprofloxicin 500mg antibiotic tablet as prophylaxis at the time of office flexible cystoscopy with ureteral stent removal. The control group will be no prophylaxis oral antibiotics. The study will be conducted at UCSD Urology outpatient clinic and Genesis Healthcare Partners Urology outpatient clinic. UCSD will be the coordinating institution.

Treatment Assignment:

Patients will be assigned to control or intervention arm based on a predetermined allocation sequence that will be generated by a computerized random number generator. Study staff not participating in patient recruitment or procedure will manage the allocation sequence. Physicians involved in urologic patient care will be blinded from the participants' allocation. Only study staff at the coordinating institution (UCSD) will have access to the full allocation sequence. i.e. no clinical staff involved in recruiting and consenting patients for the study at UCSD or other participating institutions will have knowledge of the allocation sequence at their institution prior to enrollment of each patient. To further aid allocation concealment, the block size will be varied.

Standard of care procedures:

Patients will be identified at the time of clinic visit for cystoscopic stent removal. All patients will be counseled on the American Urological Association's clinical guidelines for prophylactic antibiotic use, and the varied standardization of practice patterns. We will not deviate from routine care standards. Patients undergoing routine ureteral stent removal within two weeks following stone treatment procedure (ie. Percutaneous Nephrolithotomy, Ureteroscopy, Retrograde Intrarenal Surgery, or Extracorporal Shockwave Lithotripsy). Patients that agree to participate and provide consent will be enrolled into the study, receiving a randomized allocation, and specific data points will be collected prospectively. Patients will be consented prior to determination of prophylaxis for collection of demographic, disease, perioperative, and postoperative data. If the patient does not consent to the study the use of antibiotics will be based on the routine clinical practice of the treating urologist.

Investigational portion of treatment:

Patients randomized to the intervention arm will be provided a single oral dose of Ciprofloxacin 500mg at the time of stent removal. Ciprofloxacin is currently indicated for the treatment of acute uncomplicated urinary tract infections. Patients with fluoroquinalone allergy will receive Bactrim (trimethoprim/sulfamethoxazole 160/800mg) single dose instead of Ciprofloxacin. Those patients that do develop infectious complications after stent removal will be treated empirically based on the preference of the treating physician followed by culture specific antibiotics. Centeral prophylaxis randomization will take place at UCSD, as the lead site, using staff members not involved in patient management. Randomization will occur in block randomization in block sizes of 10.

Standard of care procedures Patients will have cystoscopy and stent removal performed in standard fashion, without deviation from standard of care. The time frame of stent removal after initial stone procedure is consistent with current standard of care. If the treating physician's preference is to maintain the patient's indwelling stent for longer than two weeks, then the patient would not be considered for this study. No patient's management course will be altered for inclusion into this study.

All female patients are screened with a urinary pregnancy test during the preoperative screening visit, which occurs before the kidney stone surgery. Any pregnant female patients will be excluded from participation in this study. Post-operative instructions include refraining from sexual activity. Cystoscopic stent removal is performed within 14 days of surgery.

Demographic fields that will be obtained preoperatively include age, race, gender, body mass index (BMI), and comorbidities including history of diabetes mellitus, immunosuppression, prior urinary tract infection(s), neurogenic bladder, incomplete bladder emptying. Pre-operative clinical data points will include kidney stone size (largest diameter as measured on coronal imaging for either kidney-ureter-bladder plain x-ray or computerized tomography) and pre-operative urine culture results.

Post-procedure fields will include post-void residual urine volume per bladder scan (to assess emptying capability), culture of urine collected during stent removal (only to be treated with antibiotics if patient becomes symptomatic - per standard of care), stone culture results, stone analysis, and stone-free status. Phone call interview will occur between 7-14 days post-operatively to determine if any post-operative infectious events have occurred. Any infectious symptoms (see below) will prompt mid-stream clean catch specimen for urinalysis and urine culture. During this period, patients will be closely observed for infectious complication--ie. symptomatic urinary tract infection, defined as presence of bacteruria (>5k colony forming units) with any of the following: fever >38 C, malodorous urine, dysuria, urinary frequency, urinary urgency, lower abdominal discomfort, back pain, gross hematuria. . Patients will be evaluated at 8 weeks for re-assessment in the clinic with a renal bladder ultrasound performed at 6 weeks, which is the routine post-operative care.

ELIGIBILITY:
Age: >=18 years of age

Gender: both men and women included. We anticipated enrolling a study population of approximately 60% men and 40% women based on a higher incidence of kidney stones among men in NHANES data.

Ethnic background: all ethnicities will be included in the study population and the specific ethnic diversity present in the study population will reflect the geographic distributions of the participating institutions.

Health Status: see below for specific inclusion/exclusion criteria.

Inclusion criteria:

* Patients with indwelling ureteral stents placed within the 2 weeks prior to the procedure visit for removal
* Patients having underwent kidney stone treatment surgery (shockwave lithotripsy [SWL], ureteroscopy [URS], retrograde intrarenal surgery [RIRS], percutaneous nephrolithotomy [PNL]) Exclusion criteria
* Patients with indwelling urethral catheter
* Patients with indwelling suprapubic catheter
* Patients with indwelling nephrostomy tube
* Patients who perform clean intermittent catheterization
* Pregnancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-01; Primary Completion 2025-01 (Actual); Study Completion 2025-03 (Actual)

PRIMARY OUTCOMES:
Post-procedure Infectious Complication | 30 days
  Urinary Tract Infection (UTI)

SECONDARY OUTCOMES:
Patient Risk Factors Predisposing to Post-procedure Infectious Complications | 30 days
  Urinary Tract Infection (UTI) Risk Factors

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Secure Server Data Sharing System

REFERENCES:
- [Background] National Nosocomial Infections Surveillance (NNIS) report, data summary from October 1986-April 1996, issued May 1996. A report from the National Nosocomial Infections Surveillance (NNIS) System. Am J Infect Control. 1996 Oct;24(5):380-8. No abstract available. PMID 8902113
- [Background] Urban JA. Cost analysis of surgical site infections. Surg Infect (Larchmt). 2006;7 Suppl 1:S19-22. doi: 10.1089/sur.2006.7.s1-19. PMID 16834543
- [Background] Wolf JS Jr, Bennett CJ, Dmochowski RR, Hollenbeck BK, Pearle MS, Schaeffer AJ; Urologic Surgery Antimicrobial Prophylaxis Best Practice Policy Panel. Best practice policy statement on urologic surgery antimicrobial prophylaxis. J Urol. 2008 Apr;179(4):1379-90. doi: 10.1016/j.juro.2008.01.068. Epub 2008 Feb 20. PMID 18280509
- [Background] Ramaswamy K, Shah O. Antibiotic prophylaxis after uncomplicated ureteroscopic stone treatment: is there a difference? J Endourol. 2012 Feb;26(2):122-5. doi: 10.1089/end.2011.0360. Epub 2011 Oct 17. PMID 22003847